CLINICAL TRIAL: NCT07357649
Title: Prospective Evaluation of Baricitinib's Effects on Procoagulant State and Atherogenic Index in Rheumatoid Arthritis Patients
Brief Title: Baricitinib Effects on Procoagulant State in Rheumatoid Arthritis
Acronym: BAR-RA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nourhan Elsaeed Abdelmabod Elhaish, Principal Investigator, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAR-RA-TANTA-2025
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental)
  Interventions: Drug: Baricitinib
- Conventional DMARD therapy (No Intervention)

INTERVENTIONS:
Drug: Baricitinib — Oral baricitinib administered in combination with methotrexate according to standard clinical practice
  Arms: Baricitinib

SUMMARY:
This prospective interventional study aims to evaluate the effects of baricitinib on disease activity, lipid profile, atherogenic index, and procoagulant biomarkers including monocyte-derived human tissue factor and D-dimer in patients with rheumatoid arthritis, compared with conventional therapy.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic systemic inflammatory disease associated with increased cardiovascular and thrombotic risk. Baricitinib, a Janus kinase 1 and 2 inhibitor, is approved for the treatment of moderate to severe rheumatoid arthritis; however, concerns remain regarding its potential prothrombotic effects.

In this prospective study, patients with rheumatoid arthritis will be recruited from Tanta University Hospitals and allocated into two parallel groups. The intervention group will receive baricitinib in combination with methotrexate after failure of conventional therapy, while the control group will continue conventional treatment.

Clinical assessment, disease activity score (DAS28), functional status (MHAQ), lipid profile, atherogenic index, monocyte-derived human tissue factor, and D-dimer levels will be evaluated at baseline and after three months to assess thrombotic risk and cardiovascular safety.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years.
* Diagnosis of rheumatoid arthritis according to the ACR/EULAR 2010 criteria.
* Patients with active rheumatoid arthritis despite conventional treatment.
* Ability to provide written informed consent.

Exclusion Criteria:

* Presence of other autoimmune diseases.
* Diabetes mellitus.
* Dyslipidemia or use of lipid-lowering therapy within the last 6 months.
* Chronic kidney disease.
* Chronic liver disease.
* Chronic respiratory disease.
* History of malignancy.
* Pregnancy or breastfeeding.
* Alcohol or drug abuse.
* Acute or chronic infection.
* Current prednisone dose > 7.5 mg/day.
* History of arterial or venous thrombosis.
* Use of anticoagulant or antithrombotic drugs within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Monocyte-Derived Human Tissue Factor Level | Baseline and 3 months
  Change in tissue factor level from baseline to 3 months after initiation of baricitinib therapy.

SECONDARY OUTCOMES:
Change in Disease Activity Score (DAS28) | Baseline and 3 months
  Change in DAS28 from baseline to 3 months.
Change in Total Cholesterol Level | Baseline and 3 months
  Change in total cholesterol level from baseline to 3 months.
Change in Triglyceride Level | Baseline and 3 months
  Change in triglyceride level from baseline to 3 months.
Change in HDL-Cholesterol Level | Baseline and 3 months
  Change in HDL-C level from baseline to 3 months.
Change in LDL-Cholesterol Level | Baseline and 3 months
  Change in LDL-C level from baseline to 3 months
Change in Atherogenic Index (TC/HDL-C) | Baseline and 3 months
  Change in atherogenic index from baseline to 3 months.
Change in D-dimer Level | Baseline and 3 months
  Change in D-dimer level from baseline to 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No